CLINICAL TRIAL: NCT00727883
Title: Retrospective Observational Trial on Reasons for Withdraw of Adjuvant Tamoxifen in Breast Cancer Patients
Acronym: SOSTA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Davide Meani Specialty Medical Affairs Manager, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-OIT-DUM-2006/1
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Adjuvant TAM; post-menopausal; women
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Post menopausal women treated with adjuvant TAM for breast cancer

SUMMARY:
Retrospective observational trial on reasons for withdraw of Adjuvant Tamoxifen in Breast Cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Breast Ca Patients with surgery and withdraw of adjuvant treatment with Tamoxifen for Tam related AEs
* Documented reasons for treatment withdrawal

Exclusion Criteria:

* enrollment in other studies
* treatment withdraw for other causes than Tam related AEs

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Post menopausal women treated with adjuvant TAM for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
incidence of withdraw from adjuvant Tamoxifen due to Tam related AEs | January 2003-December 2004

SECONDARY OUTCOMES:
Types of TAM related AE | January 2003-December 2004